CLINICAL TRIAL: NCT00291135
Title: Study of the Effect of Letrozole on Breast Biomarkers of High Risk Postmenopausal Women Receiving Hormone Replacement Therapy
Brief Title: Protocol for Women at Increased Risk of Developing Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carol Fabian, MD (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 8884
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: breast atypia; open label pilot study; letrozole; fine needle aspiration; high risk for breast cancer; breast epithelial hyperplasia; Ki-67; hormones plus chemoprevention; chemoprevention
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Oral Letrozole 2.5 mg daily for six months
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: letrozole — Letrozole 2.5 mg daily
  Other Names: Femara

SUMMARY:
A pilot study to assess the effects of six months of letrozole on breast tissue risk markers in postmenopausal women on hormone replacement therapy at high risk of developing breast cancer.

DETAILED DESCRIPTION:
A pilot study of letrozole in postmenopausal women on hormone replacement therapy at high risk of developing breast cancer. Subjects will have hyperplasia with atypia (or borderline Epithelial Hyperplasia/Atypical Hyperplasia) and evidence of Estrogen Receptor expression by random periareolar fine needle aspiration and baseline serum estradiol levels less than or equal to 150 pg/ml. The feasibility of performing RT-qPCR on breast specimens for aromatase expression will also be done at baseline.

ELIGIBILITY:
Inclusion Criteria:

* evidence of hyperplasia with/without atypia upon random periareolar fine needle aspiration of breast
* on hormone replacement therapy
* postmenopausal
* increased risk of developing breast cancer based on personal or family history
* never have taken aromatase inhibitors or selective estrogen receptor modulators in last six months
* women who have a high risk of breast cancer
* older than 18 years

Exclusion Criteria:

* anticoagulants
* marked breast tenderness
* pregnant or within twelve months of breast feeding/childbirth

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Global results will be published.

REFERENCES:
- [Background] Frank DH, Kimler BF, Fabian CJ, Ranger-Moore J, Yozwiak M, Bartels HG, Alberts DS, Bartels PH. Digital image analysis of breast epithelial cells collected by random periareolar fine-needle aspirates (RPFNA) from women at high risk for breast cancer taking hormone replacement and the aromatase inhibitor, letrozole, for six months. Breast Cancer Res Treat. 2009 Jun;115(3):661-8. doi: 10.1007/s10549-008-0274-0. Epub 2009 Jan 6. PMID 19125322
- [Result] Fabian CJ, Kimler BF, Zalles CM, Khan QJ, Mayo MS, Phillips TA, Simonsen M, Metheny T, Petroff BK. Reduction in proliferation with six months of letrozole in women on hormone replacement therapy. Breast Cancer Res Treat. 2007 Nov;106(1):75-84. doi: 10.1007/s10549-006-9476-5. Epub 2007 Jan 13. PMID 17221152
- [Result] Bartels PH, Fabian CJ, Kimler BF, Ranger-Moore JR, Frank DH, Yozwiak ML, Alberts DS. Karyometry of breast epithelial cells acquired by random periareolar fine needle aspiration in women at high risk for breast cancer. Anal Quant Cytol Histol. 2007 Apr;29(2):63-70. PMID 17484269

RESULTS

PARTICIPANT FLOW:
Groups:
- Letrozole: Letrozole, 2.5 mg daily for six months
Period: Overall Study
Arm/Group | Letrozole
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Letrozole
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Proliferation of Breast Epithelial Cells Obtained by Random Periareolar Fine Needle Aspiration.
Description: Proliferation assessment by immunocytochemistry using Ki-67. Expressed as percent of cells staining positive for Ki-67.
Time Frame: Baseline, 6 months
Population: All subjects completed study and were used for analysis
Measure: Median (Full Range); unit: Change in % of cells positive for Ki-67
Arm/Group | Letrozole
Number analyzed (Participants) | 42
Change in % of cells positive for Ki-67 | -2.3 [-21.0 to 7.8]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Letrozole
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 42/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole (N=42)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (21)
Hot Flash (Reproductive system and breast disorders) | 26 (26)
Fatigue (General disorders) | 20 (20)
alopecia (Skin and subcutaneous tissue disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes